CLINICAL TRIAL: NCT00005529
Title: Self-Scored Cardiovascular Disease Risk Appraisal
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 5062; R44HL053166 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2001-11

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Coronary Heart Disease Risk Reduction
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases

SUMMARY:
To develop and test a self-scored cardiovascular disease health risk appraisal.

DETAILED DESCRIPTION:
BACKGROUND:

Health risk appraisals (HRA) are being used increasingly by health centers and worksites to inform people of their personal mortality and morbidity risks. However, recent research suggests that many HRAs have limited reliability and validity with respect to coronary heart disease, the leading cause of death in this country. Self-scored HRAs appear to be considerably less accurate in predicting CHD risk than computerized instruments, chiefly because people do not always know the physiologic values required by these instruments and because they frequently make errors computing their scores.

DESIGN NARRATIVE:

During Phase I, a new appraisal named CardioRisk was developed. The Phase I prototype version contained eight major self-reported risk factors. CardioRisk predicted the risk of developing cardiovascular disease (CVD) in a 12-year period using an equation based on recent accelerated failure time models from the Framingham Heart Study. The purpose of Phase II was to thoroughly test and refine the prototype instrument. The Phase II analyses were designed to assess the psychometric properties of CardioRisk, to evaluate its utility as judged by patients, and to determine whether the instrument changed perceptions of personal CVD risk. These results were compared to data for other appraisals to determine whether CardioRisk outperformed comparable products.

In the proposed commercial application, CardioRisk would be distributed by health promotion organizations to increase awareness of the risk factors for cardiovascular disease. Estimates from the American Heart Association put the demand for these products at 180,000 HRAs per year. The potential market for this product includes worksites, community health centers, managed health care organizations, public health departments, and clinics.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1995-09; Study Completion 2000-08 (Actual)